CLINICAL TRIAL: NCT00336362
Title: A Pilot Study to Assess the Safety and Efficacy of G-CSF Mobilization With and Without Hydroxyurea Pretreatment in Adults With Beta Thalassemia Major
Brief Title: Evaluating the Safety of G-CSF Mobilization in Individuals With Beta Thalassemia Major
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); George Papanicolaou Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 464; 2U01HL066947 (NIH); IRB no. 27527; EudraCT no. 2005-000315-10
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Beta-Thalassemia
Keywords: Beta Thalassemia Major; Hematopoietic Stem Cell Mobilization; Gene Transfer Techniques
MeSH Terms: conditions — beta-Thalassemia | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive hydroxyurea pretreatment.
  Interventions: Drug: Hydroxyurea
- 2 (No Intervention): Participants will not receive hydroxyurea pretreatment.

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea: Subjects will be treated for one month with hydroxyurea at a starting dose of 10 mg/kg orally (closest approximation to 500 mg capsule, alternate day dosing, e.g. 500 alternating with 1000 to achieve 750 mg average daily dose), once daily, with a gradual dose escalation up to 20 mg/kg (in non-splenectomized patients) and up to 25 mg/kg (in splenectomized patients).
  G-CSF: G-CSF will be administered subcutaneously. In general, G-CSF will be administered at 10μg/kg/day (5μg/kg on a twice a day schedule) for at least 4-5 days before leukapheresis and for 1-2 additional days during collections. For the splenectomized patients who are not receiving HU pretreatment, and for the splenectomized patients who receive HU pretreatment who have greater than or equal to 12,000 WBCs before G-CSF, G-CSF will start at a lower dose (for example, 1.5 or 2.5 µg/kg); the next doses will be adjusted by the Principal Investigator based on the observed degree of leukocytosis.
  Other Names: hydrea
  Arms: 1

SUMMARY:
Beta thalassemia major is a serious genetic disease of the blood. Treatments are limited, and although a bone marrow transplant from a compatible donor can be curative, only a limited percentage of individuals with this disease have a matched donor available. A long-term goal of study researchers is to develop a gene transfer process as a method of curing beta thalassemia major. Gene transfer involves obtaining blood stem cells from an individual, adding a normal globin gene to the stem cells, and putting the cells back into the individual.

Before gene transfer methods can be attempted in individuals with beta thalassemia major, a safe method of obtaining blood stem cells needs to be developed. The purpose of this study is to investigate the safety and feasibility of collecting peripheral blood stem cells (PBSC) from individuals with beta thalassemia major. Research participants will be given G-CSF (filgrastim) for several days to increase the number of stem cells in the blood, a process called "mobilization." After mobilization, participants will undergo a procedure called apheresis to remove the white blood cells. Researchers in the laboratory will purify the stem cells from the mixture and test methods of putting a normal globin gene into the stem cells. Half of the participants will receive hydroxyurea (HU) prior to G-CSF mobilization. HU is used in splenectomized patients to attempt to reduce the risk of clotting during mobilization. In non-splenectomized patients, HU is given in an attempt to decrease the size of the spleen.

DETAILED DESCRIPTION:
Primary Objective: To determine the safety of PBSC mobilization with G-CSF, with or without HU pretreatment in adults with beta thalassemia major.

Secondary Objective: To determine the number of CD34+ stem/progenitor cells that are mobilized under these conditions, as well as the ability of these cells to be transduced with a recombinant lentivirus vector for beta-globin and engraft immunodeficient mice.

Study Design: The ability of G-CSF to safely and effectively mobilize PBSC in adults with beta thalassemia major will be assessed in 12 splenectomized and 12 non-splenectomized patients. Of the 12 splenectomized patients, 6 will be treated with HU and G-CSF, and 6 will be treated only with G-CSF. Likewise, of the 12 non-splenectomized patients, 6 will be treated with HU and G-CSF, and 6 will be treated only with G-CSF. G-CSF mobilized participants will undergo leukapheresis on 2 consecutive days, with a target yield of 2 million CD34+ cells per kg of body weight. Safety will be assessed by monitoring for study-related toxicity. Efficacy will be assessed by measuring the total number of CD34+ cells, the ability of these cells to be transduced with a recombinant lentivirus vector for beta-globin, and the ability of these cells to engraft immunodeficient mice.

Population: Adults with beta thalassemia major.

Sample size: A total of 24 subjects will be enrolled: 12 splenectomized participants and 12 non-splenectomized participants.

End Points: This is a pilot study and no specific hypotheses are being tested. However, the study will allow for qualitative comparisons if outcomes between the various arms are markedly different. For example, the study will provide qualitative data on the safety and feasibility of utilizing HU and G-CSF to mobilize stem cells in individuals with beta thalassemia major. The study will be completed upon full enrollment, or when stopping criteria are met within specific study arms.

ELIGIBILITY:
Inclusion Criteria:

* β-thalassemia major
* Karnofsky performance status greater than or equal to 80%
* Splenectomized patients or patients with spleen volume less than 800 cm^3 (V=0.523 x length x thickness x width)
* Compliant with regular transfusions and regular chelation
* Liver iron by magnetic resonance imaging (MRI) less than 280 μmol/gr or greater than or equal to 1.7 msec by T2*MRI
* Heart iron by MRI greater than 2.8 (SI/SD)or greater than or equal to 9 msec by T2*MRI
* Hepatitis B or C virus load negative by polymerase chain reaction (PCR)
* Left ventricular ejection fraction (LVEF) greater than 45% by echocardiogram or multiple gated acquisition scan (MUGA)
* Adequate respiratory function with diffusing capacity of the lung for carbon monoxide (DLCO) greater than 50%
* Negative pregnancy test, if female
* Ability to give informed consent and willingness to meet all the expected requirements of the protocol for the duration of the study

Exclusion Criteria:

* History of thrombosis or known thrombophilia
* Symptomatic viral, bacterial, or fungal infection within 6 weeks of eligibility evaluation
* Pregnant or breastfeeding
* HIV positivity
* History of cancer, other than local skin cancer
* Other systematic disease
* Splenectomized patients with platelet count greater than 900,000
* Additional risk factors for thrombosis, including Factor V Leiden; antiphospholipid antibodies; and less than 50% of the lowest normal value for the following procoagulants: antithrombin 3, protein C, or protein S

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety of PBSC mobilization with G-CSF with or without hydroxyurea pretreatment in adults with beta thalassemia major | Measured at Month 2

SECONDARY OUTCOMES:
Number of CD34+ stem/progenitor cells that are mobilized | Measured at Month 2
Ability of the obtained stem cells to be transduced with a recombinant lentivirus vector for beta-globin and engraft immunodeficient mice | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: George Stamatoyannopoulos, MD, DrSci, Study Director — University of Washington
Locations (1):
- George Papanicolaou Hospital, Thessaloniki, Greece